CLINICAL TRIAL: NCT05335434
Title: A Single Center Pilot Study of Intraoral Photobiomodulation Therapy for the Prevention of Oral Mucositis in Patients Undergoing Myeloablative Allogeneic Hematopoietic Cell Transplantation
Brief Title: Intraoral Photobiomodulation Therapy to Prevent Oral Mucositis in Patients Undergoing Hematopoietic Cell Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: THOR Photomedicine Ltd (Unknown)
Responsible Party: Principal Investigator, Kentaro Ikeda, DDS, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-036
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Myeloablative Allogeneic Hematopoietic Cell Transplantation; Intraoral Photobiomodulation Therapy; Oral Mucositis; Mucosal Ulcer
Keywords: Myeloablative Allogeneic Hematopoietic Cell Transplantation (HCT); Intraoral Photobiomodulation Therapy; Oral Mucositis; Mucosal Ulcer
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- INTRAORAL PBMT IN PATIENTS UNDERGOING alloHCT (Experimental): The research study procedures include: screening for eligibility and study treatment including daily PBMT and clinical evaluations. Participants will receive the study treatment daily from the start of conditioning chemotherapy to day +20, or discharge (if you are able to be discharged from the hospital prior to day +20), whichever occurs first
  -THOR LX2.3 with LED Lollipop
  Interventions: Device: THOR LX2.3 with LED Lollipop

INTERVENTIONS:
Device: THOR LX2.3 with LED Lollipop — The intraoral PBMT device will be placed inside of the mouth to deliver the therapeutic light. Each treatment is approximately 2-3 minutes in duration. PBMT will be administered daily starting from the start of conditioning through day +20, or discharge if prior to day +20, with 27 consecutive days defined as a maximum PBMT treatment duration

SUMMARY:
This is a single center pilot study evaluating intraoral photobiomodulation for the prevention of oral mucositis in patients undergoing myeloablative allogeneic hematopoietic cell transplantation (alloHCT). Patients who are planned for alloHCT will receive daily intraoral photobiomodulation therapy (PBMT) using a novel LED device.

The name of the study device involved in this study is:

- THOR LX2.3 with LED Lollipop

DETAILED DESCRIPTION:
As part of a transplant procedure patients will receive chemotherapy in a conditioning regimen in preparation of alloHCT as well as immunosuppressive medications to help prevent graft-versus-host disease ("GVHD prophylaxis"). Together, these treatments will put patients at risk for developing side effects. A common side effect is oral mucositis (OM), in which mouth sores develop making eating and speaking difficult and painful.

Photobiomodulation therapy (PBMT) is a light-based therapy that reduces inflammation and enhances wound healing. PBMT delivered inside the mouth has been shown to reduce OM in patients undergoing alloHCT.

The name of the study device involved in this study is:

- THOR LX2.3 with LED Lollipop

This research study is a Pilot Study, which is the first time that investigators are examining this LED based intraoral PBMT.

The U.S. Food and Drug Administration (FDA) has not approved PBMT for this specific disease but it has been approved for other uses.

The research study procedures include: screening for eligibility and study treatment including daily PBMT and clinical evaluations.

Participants will receive study treatment daily from the start of conditioning chemotherapy to day +20, or discharge (if you are able to be discharged from the hospital prior to day +20), whichever occurs first.

It is expected that about 20 people will take part in this research study

ELIGIBILITY:
Inclusion Criteria:

* Planned to undergo myeloablative allogeneic HCT using FluBu4 conditioning and Tac-Mtx GVHD prophylaxis.
* Age ≥18 years.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had treatment with intraoral PBMT within four weeks of admission for HSCT.
* Participants who have a history of radiation therapy to the head and neck.
* Participants who have a history of photosensitivity or underlying disease with known photosensitivity.
* Participants who are planned to receive palifermin for OM prevention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
Duration of severe Oral Mucositis | 20 Days
  Defined as the total number of days between day 0 and day +20 on which severe (WHO grade 3 or 4) OM was reported

CONTACTS AND LOCATIONS:
Overall Officials: Kentaro Ikeda, DDS, MPH, Principal Investigator — Brigham and Women's Hospital; Nathaniel S. Treister, DMD, DMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation